CLINICAL TRIAL: NCT06627686
Title: Predictive Value of Airway Occlusion Pressure, Maximal Inspiratory Pressure and Their Ratio for Successful Extubation in Patients With Traumatic Brain Injury Observational Study
Brief Title: Predictive Value of Airway Occlusion Pressure, Maximal Inspiratory Pressure and Their Ratio for Successful Extubation in Patients With Traumatic Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Benha University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Ali Rashad Ahmed Abd El Bary, Principal investigator, Benha University
Other Study IDs: MS 23_7_2023
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Weaning Failure
MeSH Terms: interventions — Maximal Respiratory Pressures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Traumatic brain injury: Air way occlusion pressure and maximum inspiratory pressure
  Interventions: Diagnostic Test: Air way occlusion pressure

INTERVENTIONS:
Diagnostic Test: Air way occlusion pressure — Predictive Value of Airway Occlusion Pressure, Maximal Inspiratory Pressure and Their Ratio for Successful Extubation in Patients with Traumatic Brain Injury
  Other Names: Maximal inspiratory pressure

SUMMARY:
The aim of this study will be to measure the predictive power of the respiratory muscle determinants including The maximal inspiratory pressure, and central drive determinant including Airway occlusion pressure and ratio between them in weaning outcome of traumatic brain injury patients undergoing invasive mechanical ventilation.

DETAILED DESCRIPTION:
Before spontaneous breathing trials with a T-piece for 30 min with an FIO2 of 0.40, measurements will be performed for a 20-second period. Three parameters will be analyzed: PImax, P0.1, and P0.1/PImax. PImax and P0.1 will be obtained using a unidirectional valve method and a manovacuometer (Instrumentation Industries, Bethel Park, PA) attached to the airway.

The device will have a scale of 30 cm H2O with a 1 cm H2O interval, and will be designed to perform measurements at each 0.1 second. Prior to testing, all subjects will be on pressure support ventilation mode (12-20 cm H2O) and will not be on sedatives. The head of the subject's bed will be elevated to 45 degrees and the cuff of the artificial airway will be hyperinflated to prevent air leakage during measurement.

The subject will have the airway clear of secretions by suctioning with standard tracheal suction procedures after pre-oxygenation for 2 minutes with FIO2 of 1.0.

After a brief rest period, pre-oxygenation will be repeated. The subject will then be disconnected from mechanical ventilation and allowed to breathe spontaneously for 10 seconds before connecting the artificial airway to the manovacuometer when the subject will at functional residual capacity. The subject will continuously be monitored by pulse oximetry and electrocardiogram, and will have continual respiratory physiotherapist attention.

For the present study, respiratory drive (P0.1) will be calculated as an average of the measured inspiratory pressure 0.1 s after the initiation of the inspiration for the first 3 cycles, and P0.1/PImax as the ratio of absolute values of P0.1 and PImax. The subjects will not coached for the maneuver. Thresholds for the 3 parameters will be calculated from their respective receiver operating characteristic (ROC) curves. Values more negative than -25 cm H2Owere used to predict successful weaning.

Weaning will be considered successful if spontaneous breathing will sustained for 48 hours after withdrawal from mechanical ventilation.

The trial will stopped if at least one of the following intolerance criteria present: SaO2 less than 90% or PaO2 less than 60 mm Hg with FIO2 greater than 0.4; PaCO2 greater than mm Hg or increased by 8 mm Hg or more; arterial pH less than 7.33 or decreased by 0.07 or more; respiratory rate greater than 35 breaths/ min or increased by 50% for 5 min or longer; heart rate greater than 140 beats/min or a sustained increase or decrease in 20%; mean blood pressure greater than 130mmHg or less than 70mmHg; or presence of agitation, diaphoresis, disorientation, or depressed mental status.

The subjects who will demonstrate one of these signs during the spontaneous breathing trial or within 48 hours after the discontinuation from mechanical ventilation will be considered not weaned and will returne to ventilator support.

Before being submitted to spontaneous breathing trials (SBTs) of 2 hours patients will have the tracheal P 0.1 and the PImax measured; P 0.1/PImax ratio will then be calculated.

Traditional thresholds will be adopted for the 3 parameters. Tracheal P 0.1 will be measured in pressure support ventilation, with pressure support in 7 cm H2O and positive end expiratory pressure in 5 cm H2O. At least 3 measurements, separated by an interval of not less than 15 seconds, will be obtained, and the mean value will be used for analysis. Tracheal P 0.1 values less than 4.2 cm H2O will be used to predict successful weaning.

P 0.1/PImax ratio will be obtained through the division of tracheal P 0.1 by PImax, and because both of them, in reality, are negative pressures, the result will expressed in positive values. Values smaller than 0.14 will be used to predict successful weaning.

4- Patients who will pass SBT without deterioration will extubated and receive oxygen through Venturi mask 40%. However, SBT failure will be considered if the patient develop a decreased level of consciousness, diaphoresis, RR>35 breaths/min, hemodynamic instability (heart rate>140, systolic blood pressure>180 or <90 mmHg) or signs of increased work of breathing.

ELIGIBILITY:
Traumatic brain injury (closed type) patients who will be admitted to ICU and intubated and MV more than 24 hours will be included in this study.

Age from 18 to 65 years (male or female).

Fulfillment of Criteria of readiness for weaning off MV :

Resolution of the cause of respiratory insufficiency and MV. Stable hemodynamic profile

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Predictive Value of Airway Occlusion Pressure, Maximal Inspiratory Pressure and Their Ratio for Successful Extubation in Patients with Traumatic Brain Injury
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
Sensetivity, specifity, predictive values, and accuracy of Maximal inspiratory pressure, Airway occlusion pressure and their ratio will be determined by ROC curve. | One day

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rashad, MBBCH, Principal Investigator — Benha University
Locations (1):
- Ali Rashad Ahmed, Tanta, Mahala, Egypt

IPD SHARING:
Plan to Share IPD: No